CLINICAL TRIAL: NCT00681824
Title: An Exploratory Phase 2 Study Evaluating the Efficacy and Safety of Fibrin Sealant, Vapor Heated, Solvent/Detergent Treated (FS VH S/D) 500 S-APR for the Sealing of Dura Defect Sutures in Posterior Fossa Surgery
Brief Title: Fibrin Sealant for the Sealing of Dura Sutures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 550701
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2013-06-27 (Estimated); Status verified 2013-05

CONDITIONS: Pathological Processes in the Posterior Fossa; Dura Defects
MeSH Terms: interventions — Fibrin Tissue Adhesive; Solvents; Thrombin; Low Density Lipoprotein Receptor-Related Protein-1; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- FS VH S/D 500 s-apr (Experimental): Application of FS VH S/D 500 s-apr on top of suture
  Interventions: Biological: Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr)
- Standard of Care (Control group) (Active Comparator): The treatment of the control group consisted of Standard of Care (SoC) which was defined as the closure of a dura defect by suturing in a patch of autologous fascia, pericranium or suturable collagen based dura substitute.
  Interventions: Procedure: Standard of care

INTERVENTIONS:
Biological: Fibrin Sealant, Vapor Heated, Solvent/Detergent-treated with 500 IU/mL thrombin and synthetic aprotinin (FS VH S/D 500 s-apr) — Application of a thin layer of FS VH S/D 500 s-apr to the entire length of the suture loop and the adjacent area to at least 5 mm away from the suture line, including all suture holes. After application, the product is to be allowed to polymerize for 3 minutes.
  Other Names: TISSEEL; FS VH S/D 500 s-apr (a double virus-inactivated biological two-component fibrin sealant)
  Arms: FS VH S/D 500 s-apr
Procedure: Standard of care — Standard care: defined as the closure of a dura defect by suturing in a patch of autologous fascia, pericranium or suturable collagen-based dura substitute.
  Arms: Standard of Care (Control group)

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of FS VH S/D 500 s-apr, a double virus-inactivated biological two-component fibrin sealant, for use in posterior fossa surgery as an adjunct to dura and dura substitute sutures in preventing postoperative cerebrospinal fluid (CSF) leakage.

ELIGIBILITY:
Inclusion Criteria:

Preoperative Inclusion Criteria:

* Subjects undergoing elective craniotomy / craniectomy for pathological processes in the posterior fossa (such as benign and malignant tumors, vascular malformations, and Chiari 1 malformations) that result in dura defects requiring dura substitution for closure and who are able and willing to comply with the procedures required by the protocol
* Signed and dated written informed consent from the subject or from his/her legal representative prior to any study-related procedures
* Age >= 3 years, either gender

Intraoperative Inclusion Criteria:

* Surgical Wound Classification Class I and Risk Index Category (RIC) <= 2. Penetration of mastoid air cells during partial mastoidectomy is permitted and will be recorded.
* A patch of autologous fascia or pericranium or suturable collagen-based dura substitute was cut to size and then sutured into the dura defect.
* The hem of native dura exposed along and under the craniotomy edge is wide enough to facilitate suturing and to allow for sufficient surface area for adherence of the investigational product.

Exclusion Criteria:

Preoperative Exclusion Criteria:

* Female subjects who are breastfeeding, pregnant, or intend to become pregnant during the clinical study period
* Subjects with a dura lesion from a recent surgery that still has the potential for cerebrospinal fluid (CSF) leakage unless it can be expected that the lesion will be excised completely, including all old suture holes
* Chemotherapy scheduled within 7 days following surgery
* Radiation therapy to the head scheduled within 7 days following surgery
* Subjects with severely altered renal (serum creatinine > 2 mg/dL) and/or hepatic function [ALT, AST > 5 x upper limit of norm (ULN)]
* Evidence of an infection indicated by any one of the following: fever > 101°F, white blood cell (WBC) count < 3500/μL or > 13000/μL, positive blood culture, positive chest X-ray. A positive urine culture (> 10^5 colony-forming units (CFU)/mL) leads to exclusion unless acute cystitis is the sole cause. Evidence of infection along the planned surgical path. A WBC count of < 20000/μL is permitted if the patient is being treated with steroids in the absence of all the other infection parameters.
* Conditions compromising the immune system; existence of autoimmune disease
* Known hypersensitivity to aprotinin or other components of the investigational product
* Non-compliant or insufficient treatment of diabetes mellitus [glycosylated hemoglobin (HbA1c) > 7.5%]
* Hydrocephalus, except occlusive hydrocephalus caused by posterior fossa pathology to be treated
* Existing CSF (ventricular, etc.) drains. Burr holes are permitted as long as the dura remains intact. Cushing cannulation excludes the subject.
* Female subjects of childbearing potential with a positive urine or serum pregnancy test within 24 hours prior to surgery
* Participation in another clinical trial with exposure to another investigational drug or device within 30 days prior to enrollment
* Scheduled or foreseeable surgery within the follow-up period

Intraoperative Exclusion Criteria:

* Dura injury during craniotomy / craniectomy that cannot be eliminated by recreating a sufficiently wide native dura hem
* Failure to administer preoperative antibiotic prophylaxis
* Use of implants made of synthetic materials coming into direct contact with dura (e.g., polytetrafluoroethylene (PTFE) patches, shunts, ventricular and subdural drains)
* Placement of Gliadel wafers
* Chiari 1 subjects without injury to the arachnoid
* Persistent signs of increased brain turgor
* Use of product(s) other than FS VH S/D 500 s-apr for the sealing of dura sutures, including packing with Gelfoam
* Brain surface visible between suture loops as a manifestation of increased suture tension
* CSF leakage from completed dura sutures presenting as dripping drops, growing beads or running trickles. Slight oozing is consistent with successful dura repair and will not lead to exclusion.
* Intersecting durotomy scars in the surgical path from a previous operation that cannot be completely removed by the planned dura resection
* Dura lesion from a recent surgery that cannot be completely excised, including all old suture holes
* Two or more separate dura defects
* Major intraoperative complications that require resuscitation or deviation from the planned surgical procedure

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2008-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guenter Zuelow, MD, Study Director — Baxter Healthcare Corporation
Locations (13):
- United States (12):
  - Duarte, California
  - Sacramento, California
  - San Diego, California
  - Orlando, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Louisville, Kentucky
  - Johnson City, New York
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
- Hamilton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 12 United States and 1 Canadian clinical site(s) beginning May 2008 and completing in March 2010
Pre-assignment Details: 95 were enrolled. 23 discontinued (10 screen failures, 3 withdrawn by investigator, 3 withdrawn by representative or self, 1 died- failure to thrive, 1 had surgery before randomized, 1 study site distance, 1 site reached enrollment goal, 2 patients cancelled surgery, 1 family delayed >30 day window. 62 randomized. There were 13 run-in participants.
Groups:
- Standard of Care: The closure of a dura defect by suturing in a patch of autologous fascia, pericranium or suturable collagen-based dura substitute.
- Run-in Participants: FS VH S/D 500 S-apr: One initial
- FS VH S/D 500 S-apr: Application of thin layer of FS VH S/D 500 s-apr to entire length of suture loop and adjacent area to at least 5 mm away from the suture line, including all suture holes. After application, the product is to be allowed to polymerize for 3 minutes.
Period: Overall Study
Arm/Group | Standard of Care | Run-in Participants: FS VH S/D 500 S-apr | FS VH S/D 500 S-apr
Started | 28 | 13 | 34
Completed | 27 | 12 | 33
Not Completed | 1 | 1 | 1
Not completed — withdrawn by investigator | 0 | 0 | 1
Not completed — scheduling conflict | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Primary Safety Dataset Note: This includes 13 initial "run-in" participants in the FS VH S/D 500 s-apr arm (one for each site permitted to familiarize the investigators with the study procedures)
Groups:
- Standard of Care (SoC): The closure of a dura defect by suturing in a patch of autologous fascia, pericranium or suturable collagen-based dura substitute.
- FS VH S/D 500 S-apr (Run-In Participants Only): Application of thin layer of FS VH S/D 500 s-apr to entire length of suture loop and adjacent area to at least 5 mm away from the suture line, including all suture holes. After application, the product is to be allowed to polymerize for 3 minutes. Note: This arm/group only includes the 13 initial "run-in" participants (one for each site permitted to familiarize the investigators with the study procedures)
- FS VH S/D 500 S-apr (Non Run-In Participants Only): Application of thin layer of FS VH S/D 500 s-apr to entire length of suture loop and adjacent area to at least 5 mm away from the suture line, including all suture holes. After application, the product is to be allowed to polymerize for 3 minutes. Note: This arm/group does not include the 13 initial "run-in" participants (one for each site permitted to familiarize the investigators with the study procedures)
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SoC) | FS VH S/D 500 S-apr (Run-In Participants Only) | FS VH S/D 500 S-apr (Non Run-In Participants Only) | Total
Number analyzed (Participants) | 28 | 13 | 34 | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 40.2 (19.7) | 42.9 (20.34) | 33.3 (19.01) | 37.5 (19.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 21 | 48
  Male | 11 | 3 | 13 | 27
Region of Enrollment [Number; unit: participants]
  United States | 25 | 12 | 30 | 67
  Canada | 3 | 1 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Cerebrospinal Fluid (CSF) Leakage Observed After Surgery
Description: Study-relevant CSF leakage is defined as one or more of following:
  1. Discrete subcutaneous or subgaleal CSF collection (pseudomeningocele) in surgical area confirmed by positive test for β2-transferrin, or by computed tomography (CT) or magnetic resonance imaging (MRI)
  2. Epidural CSF collection in surgical area depicted by CT or MRI
  3. Leakage of CSF through surgical wound observed during physical examination, confirmed by a positive test for β2-transferrin
  4. Progressive pneumatocephalus (air in subarachnoidal space) depicted by repeat CT in absence of CSF drainage.
Time Frame: 33 +/- 3 days after surgery
Population: Intent to treat
  One participant (SoC arm) received products other than FS VH S/D 500 s-apr for sealing of dura sutures and was removed from analysis
  Two participants (FS VH S/D 500 s-apr arm) removed from analysis due to (1) subsequent surgery unrelated to CSF leakage/surgical site infection that involved re-durotomy (2) withdrew from study
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr: Application of thin layer of FS VH S/D 500 s-apr to entire length of suture loop and adjacent area to at least 5 mm away from the suture line, including all suture holes. After application, the product is to be allowed to polymerize for 3 minutes. Note: This arm/group does not include 13 initial run-in participants (one for each site permitted to familiarize the investigators with the study procedures)
Arm/Group | Standard of Care (SoC) | FS VH S/D 500 S-apr
Number analyzed (Participants) | 27 | 32
percentage of participants | 74.07 [55.32 to 86.83] | 78.13 [61.25 to 88.98]
Statistical Analysis 1: Comparison: Standard of Care (SoC) vs FS VH S/D 500 S-apr; Test type: Superiority or Other; p = 0.7159, likelihood ratio of chi squared test

2. Secondary Outcome: Incidence of Procedures Resulting From the Treatment of CSF Leaks
Description: The incidence of surgical revisions, number and duration of compression bandage applications and of liquor drainage procedures
Time Frame: until resolution or 30 days after final follow-up visit (Day 33+/-3), whichever is first
Population: Intent to treat
  One participant (SoC arm) received products other than FS VH S/D 500 s-apr for sealing of dura sutures and was removed from analysis
  One participant (FS VH S/D 500 s-apr arm) removed from analysis due to subsequent surgery unrelated to CSF leakage/surgical site infection that involved re-durotomy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care (SoC) | FS VH S/D 500 S-apr
Number analyzed (Participants) | 27 | 33
percentage of participants
  Surgical Revision | 0 [NA to NA] — There were no procedures for this group | 3.03 [0.54 to 15.32]
  Compression Bandage | 0 [NA to NA] — There were no procedures for this group | 0 [NA to NA] — There were no procedures for this group
  Liquor Drainage | 0 [NA to NA] — There were no procedures for this group | 0 [NA to NA] — There were no procedures for this group

3. Secondary Outcome: Number of Participants With Procedures Resulting From the Treatment of CSF Leaks
Description: The number of participants with surgical revisions, number and duration of compression bandage applications and of liquor drainage procedures.
Time Frame: until resolution or 30 days after final follow-up visit (Day 33+/-3), whichever is first
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Standard of Care (SoC) | FS VH S/D 500 S-apr
Number analyzed (Participants) | 27 | 33
participants
  Surgical Revision | 0 [NA to NA] | 1 [0.54 to 15.32]
  Compression Bandage | 0 [NA to NA] | 0 [NA to NA]
  Liquor Drainage | 0 [NA to NA] | 0 [NA to NA]

4. Primary Outcome: Number of Participants With Cerebrospinal Fluid (CSF) Leakage Observed After Surgery
Description: as for outcome 1
Time Frame: 33 +/- 3 days after surgery
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Standard of Care (SoC) | FS VH S/D 500 S-apr
Number analyzed (Participants) | 27 | 32
participants | 20 | 25

5. Secondary Outcome: Incidence of Surgical Site Infections (SSI) According to National Nosocomial Infection Surveillance (NNIS) Criteria
Time Frame: within 1 month following surgery
Population: Primary Safety Data Set
  One participant (FS VH S/D 500 s-apr arm) removed from analysis due to subsequent surgery unrelated to CSF leakage/surgical site infection that involved re-durotomy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- FS VH S/D 500 S-apr: Application of thin layer of FS VH S/D 500 s-apr to entire length of suture loop and adjacent area to at least 5 mm away from the suture line, including all suture holes. After application, the product is to be allowed to polymerize for 3 minutes. Note: This arm/group includes 13 initial run-in participants (one for each site permitted to familiarize the investigators with the study procedures)
Arm/Group | Standard of Care | FS VH S/D 500 S-apr
Number analyzed (Participants) | 28 | 46
percentage of participants | 0.00 [NA to NA] — There were no SSIs for this group | 2.17 [0.38 to 11.34]

6. Secondary Outcome: Number of Participants With Surgical Site Infections (SSI) According to National Nosocomial Infection Surveillance (NNIS) Criteria
Time Frame: within 1 month following surgery
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Standard of Care | FS VH S/D 500 S-apr
Number analyzed (Participants) | 28 | 46
participants | 0 [NA to NA] | 1 [0.38 to 11.34]

ADVERSE EVENTS:
Time Frame: Throughout the study period, 1 year and 10 months
Groups:
- FS VH S/D 500 S-apr: Application of thin layer of FS VH S/D 500 s-apr to entire length of suture loop and adjacent area to at least 5 mm away from the suture line, including all suture holes. After application, the product is to be allowed to polymerize for 3 minutes. Note: This arm/group includes 13 initial "run-in" participants (one for each site permitted to familiarize the investigators with the study procedures)
Arm/Group | Standard of Care (SoC) | FS VH S/D 500 S-apr
Serious Adverse Events (participants affected / at risk) | 4/28 | 10/47
Other Adverse Events (participants affected / at risk) | 20/28 | 33/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=28) | FS VH S/D 500 S-apr (N=47)
Intracranial hypotension (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pseudomeningocele (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 2 (2)
Meningitis aseptic (Nervous system disorders) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SoC) (N=28) | FS VH S/D 500 S-apr (N=47)
Diplopia (Eye disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (6) | 5 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 5 (5)
Candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3)
Incision site pain (Injury, poisoning and procedural complications) | 15 (15) | 25 (25)
Pseudomeningocele (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 4 (4)
Hypertension (Vascular disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxter's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until the earlier of the primary multicenter publication or 12 months after study completion. Baxter requires a review of results communications (e.g., for confidential information) ≥45 days prior to submission or communication. Baxter may request an additional delay of ≤60 days e.g., for intellectual property protection)